CLINICAL TRIAL: NCT02038478
Title: Nonmyeloablative Allogeneic Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation for Severe Congenital Anemias Including Sickle Cell Disease and Thalassemia
Brief Title: Allograft for Sickle Cell Disease and Thalassemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Prapti Patel, PI, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 012013-015
Record Dates: First submitted 2014-01-10; First posted 2014-01-16 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Sickle Cell Disease and Thalassemia
Keywords: Sickle Cell Disease; Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transplantation Arm (Experimental): Transplantation
  One day after they complete their radiation and Campath-1H treatments and have begun their Sirolimus, the donor blood stem cells described above are transfused through the central line. This process takes approximately 30 minutes to 2 hours and is normally completely without side effects.
  Interventions: Biological: Donor Stem Cell Transplantation

INTERVENTIONS:
Biological: Donor Stem Cell Transplantation — One day after they complete their radiation and Campath-1H treatments and have begun their Sirolimus, the donor blood stem cells described above are transfused through the central line. This process takes approximately 30 minutes to 2 hours and is normally completely without side effects.

SUMMARY:
The design of the study incorporates the following features:

1. This is a phase II study to determine the safety and therapeutic potential of a new transplant approach (disease-free survival, graft versus myeloma effect) and to evaluate its toxicity profile (immediate toxicity, graft-versus-host disease, graft rejection, mortality) in a patient population with severe congenital anemias.
2. The patient cohort to be studied: Those patients with severe sickle cell disease and thalassemia who have risk factors for high mortality and morbidity related to their disease
3. Transplant Conditioning Regimen - Immunosuppression without myeloablation: Patients will receive conditioning sufficient to allow donor lympho-hematopoietic engraftment without complete marrow ablation. If the graft is rejected, the patient will reconstitute autologous marrow function. We will use a combination of low dose irradiation, Alemtuzumab (Campath®), and sirolimus.
4. Peripheral blood hematopoietic progenitor cell (PBPC) transplant: An unmanipulated peripheral blood stem cell collection from a filgrastim (G-CSF) stimulated HLA-matched donor should improve the chance of engraftment because of the high stem cell dose (5 x 106/kg CD34+ cells) and the presence of donor lymphocytes. To reduce the risk of GVHD, patients will receive sirolimus before and after the transplant. The sirolimus will be tapered as necessary to minimize any graft versus host disease while still maintaining adequate chimerism.

DETAILED DESCRIPTION:
A human lymphocyte antigen (HLA)-matched sibling donor will receive filgrastim (G-CSF) 10 to16 µg/kg/d subcutaneously or intravenously for up to 6 days with apheresis collections of PBPC on day 5 (and day 6 if required). The product will be collected by leukophoresis with a goal of ≥ 10 x 106 CD34+ cells/kg, with a minimum of 5 x 106 CD34+ cells/kg.

The patient will receive a preparative regimen of Alemtuzumab to be infused on days -7 to -3, followed by 300 cGy TBI given as a single dose on day -2. Sirolimus at a dose of 5mg/day to maintain trough levels between 10-15ng/ml will be started on day -1. The PBPC graft targeted to deliver 10 x 106 CD34+ cells/kg (at minimum, 5 x 106 CD34+ cells/kg) will be infused on day 0 On days +14, +30, +60 and +100 the chimeric status of patients will be assessed by microsatellite analysis of the peripheral blood. More frequent monitoring may be required.

Sickle cell patients with pulmonary hypertension will meet with a Pulmonary Medicine Consult to determine appropriate management prior to SCT.

Patients with fever or suspected minor infection should await resolution of symptoms before starting the conditioning regimen.

Iron chelation must be discontinued > 48 hours before initiating the conditioning regimen.

Hydroxyurea must be discontinued one day prior to initiating the conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria - Recipient

Disease specific:

Sickle Cell Disease - Patients with sickle cell disease at high risk for disease related morbidity or mortality, defined by having irreversible end-organ damage (A, B, C,D, or E) or potentially reversible complication(s) not ameliorated by hydroxyurea (F):

A. Stroke defined as a clinically significant neurologic event that is accompanied by an infarct on cerebral MRI OR an abnormal trans-cranial Doppler examination (≥200m/s); OR

B. Sickle cell related renal insufficiency defined by a creatinine level ≥1.5 times the upper limit of normal and kidney biopsy consistent with sickle cell nephropathy OR nephrotic syndrome OR creatinine clearance < 50mL/min OR requiring peritoneal or hemodialysis. OR

C. Pulmonary hypertension as defined by tricuspid regurgitant jet velocity (TRV) of ≥ 2.5m/s at least 3 weeks after a vaso-occlusive crisis; OR

D. Recurrent tricorporal priapism defined as at least two episodes of an erection lasting ≥4 hours involving the corpora cavernosa and corpus spongiosa; OR

E. Sickle hepatopathy defined as EITHER ferritin >1000mcg/L OR direct bilirubin >0.4 mg/dL at baseline; OR

F. Any one of the below complications

1. Vaso-occlusive crises
2. Acute chest syndrome
3. Osteonecrosis of 2 or more joints
4. Red cell alloimmunization

   Thalassemia - Patients with thalassemia who have grade 2 or 3 iron overload, determined by the presence of 2 or more of the following:

   • portal fibrosis by liver biopsy inadequate chelation history (defined as failure to maintain adequate compliance with chelation with desferroxamine initiated within 18 months of the first transfusion and administered subcutaneously for 8-10 hours at least 5 days each week) hepatomegaly of greater than 2 cm below the costochondral margin

   Non-disease specific:

   Ages ≥ 18 but ≤ 45

   6/6 HLA matched family donor available

   Ability to comprehend and willing to sign an informed consent, assent obtained from minors

   Negative serum pregnancy test

   Inclusion criteria - Donor

   6/6 HLA identical family donor

   Weight > 20 kg (in so far that the weight difference between recipient and donor does not exceed a reasonable likelihood of being able to obtain an adequate cell dose from the donor within two aphereses)

   Fit to receive G-CSF and give peripheral blood stem cells (normal blood counts, normotensive, and no history of stroke)

   Ability to comprehend and willing to sign an informed consent

   Exclusion Criteria:

   Exclusion criteria - Recipient

   Any of the following would exclude the subject from participating

   ECOG performance status of 3 or more or Lanksy performance status of <40

   Diffusion capacity of carbon monoxide (DLCO) <50% predicted (corrected for hemoglobin and alveolar volume)

   Baseline oxygen saturation of <85% or PaO2 <70

   Left ventricular ejection fraction: <40% estimated by ECHO

   Transaminases > 5x upper limit of normal for age

   Evidence of uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms) within one month prior to starting the conditioning regimen

   Major anticipated illness or organ failure incompatible with survival from PBSC transplant

   Pregnant or lactating

   Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

   Major ABO mismatch

   Exclusion criteria - Donor

   Any of the following would exclude the donor from participating

   Pregnant or lactating

   Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)

   HIV positive

   Hemoglobin S > 50%, or beta thalassemia intermediate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2021-01 (Estimated); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Treatment Success at One Year | Treatment Success at one year
  This is defined as full donor type hemoglobin on hemoglobin electrrophoresis for patients with sickle cell disease and transfusion-independence for patients with thalassemia.

SECONDARY OUTCOMES:
Level of chierism required to maintain Graft Survival and hematologic normalcy | Measured on days 14, 30, 60 and 100
  The chimeric status of patients will be measured on days +14, +30, +60, and +100 by microsatellite analysis of the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Prapti Patel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States